CLINICAL TRIAL: NCT03534453
Title: An Open Label, Single Arm, Multicentre Study to Assess the Clinical Efficacy and Safety of Lynparza (Olaparib) Tablets Maintenance Monotherapy in Platinum Sensitive Relapsed Ovarian Cancer Patients Who Are in Complete or Partial Response Following Platinum Based Chemotherapy (L-MOCA)
Brief Title: Olaparib Tablets Maintenance Monotherapy Ovarian Cancer Patients After Complete or Partial Response to Platinum Chemotherapy
Acronym: L-MOCA
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: D0816C00016
Record Dates: First submitted 2018-03-12; First posted 2018-05-23 (Actual); Last update posted 2025-07-10 (Actual); Status verified 2025-07

CONDITIONS: Relapsed Ovarian Cancer; Following Complete or Partial Response to Platinum Based Chemotherapy; Platinum Sensitive
Keywords: ovarian cancer; PARP Inhibitor; Platinum sensitive
MeSH Terms: conditions — Ovarian Neoplasms | interventions — olaparib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Olaparib 300mg tablets (Experimental): Taken orally twice daily
  Interventions: Drug: Olaparib 300mg tablets

INTERVENTIONS:
Drug: Olaparib 300mg tablets — 300mg Olaparib tablets taken orally twice daily until objective radiological disease progression as per RECIST as assessed by the investigator (or as long as in the investigator's opinion they are benefiting from treatment and they do not meet any other discontinuation criteria). Dose reduction to 250mg and subsequently 200mg is permitted following confirmation of toxicity.

SUMMARY:
This is a prospective, open-label, single arm, multi-centre interventional study to assess the clinical efficacy and safety of olaparib maintenance monotherapy and will be conducted in patients with platinum sensitive relapsed (PSR) high grade epithelial ovarian, fallopian tube, or primary peritoneal cancer who are in response (complete response or partial response) to platinum-based chemotherapy

DETAILED DESCRIPTION:
Eligible patients will be those with high grade (serous or endometrioid) epithelial ovarian cancer, primary peritoneal and/or fallopian tube cancer.

Patients must have completed 2 previous lines of platinum-based therapy (e.g., containing carboplatin or cisplatin) and platinum sensitive relapsed before entry to the study. Eligible patients must be in complete or partial response according to RECIST 1.1 criteria following the platinum-based chemotherapy prior to enrolment in the study.

BRCA (Breast Cancer Susceptibility genes) and HRR (Homologous Recombination Repair) mutation status should be determined through blood and/or tumour testing when patients are enrolled in this study.

Patients will be assigned olaparib tablets p.o. 300 mg twice daily. They should initiate olaparib treatment within 8 weeks after their last dose of platinum-containing chemotherapy (last dose is the day of the last infusion).

Patients must have clinical and objective radiological tumour assessments according to Response Evaluation Criteria in Solid Tumors (RECIST 1.1) criteria at baseline and every 12 weeks relative to date of enrolment, until objective radiological disease progression as determined by the investigator. Patients could continue to receive olaparib for as long as determined by the investigator, until objective radiological disease progression or as long as in the investigator's opinion they are benefiting from treatment in relation to other clinical assessments and they do not meet any other discontinuation criteria. Once a patient has discontinued olaparib she will be managed as per local clinical practice but will remain in the study and data will be collected on subsequent treatments, progression, overall survival and safety.

ELIGIBILITY:
Inclusion Criteria:

1. Provision of informed consent prior to any study specific procedures
2. Age 18 years or over
3. Patients with platinum sensitive relapsed high grade (serous or endometrioid) epithelial ovarian cancers (including primary peritoneal and/or fallopian tube cancer)

   * Platinum sensitive disease is defined as disease progression ≥6 months after completion of their last dose of platinum based chemotherapy
4. Patients should have received at least 2 previous lines of platinum containing therapy prior to enrolment:

   * For the last chemotherapy course immediately prior to enrolment on the study, patients must be, in the opinion of the investigator, in response (partial or complete radiological response according to RECIST 1.1 criteria) and no evidence of a rising CA-125, following completion of this chemotherapy course.
5. Have availability of 10 ml blood for germline BRCA testing and tumor sample for sBRCA and HRRm testing: paraffin-embedded archived tumor tissue block (preferred) or, if a block is not possible, it would be better to have qualified 15 5-μm unstained sections.
6. Patients must have normal organ and bone marrow function measured within 28 days prior to administration of study treatment as defined below:

   * Haemoglobin ≥ 10.0 g/dL with no blood transfusions in the past 28 days
   * Absolute neutrophil count (ANC) ≥ 1.5 x 109/L
   * Platelet count ≥ 100 x 109/L
   * Total bilirubin ≤ 1.5 x institutional upper limit of normal (ULN)
   * Aspartate aminotransferase (AST) (Serum Glutamic Oxaloacetic Transaminase (SGOT)) / Alanine aminotransferase (ALT) (Serum Glutamic Pyruvate Transaminase (SGPT)) ≤ 2.5 x institutional upper limit of normal unless liver metastases are present in which case they must be ≤ 5x ULN
   * Patients must have creatinine clearance estimated using the Cockcroft-Gault equation of ≥51 mL/min:

   Estimated creatinine clearance =[(140-age [years]) x weight (kg)]/[serum creatinine (mg/dL) x 72] (x F)a

   a: where F=0.85 for females and F=1 for males.
7. Eastern Cooperative Oncology Group (ECOG) performance status 0-1.
8. Patients must have a life expectancy ≥ 16 weeks.
9. Postmenopausal or evidence of non-childbearing status for women of childbearing potential: negative urine or serum pregnancy test within 28 days of study treatment and confirmed prior to treatment on day 1.

   Postmenopausal is defined as:
   * Amenorrheic for 1 year or more following cessation of exogenous hormonal treatments
   * Luteinizing hormone (LH) and Follicle stimulating hormone (FSH) levels in the post menopausal range for women under 50
   * radiation-induced oophorectomy with last menses >1 year ago
   * chemotherapy-induced menopause with >1 year interval since last menses
   * surgical sterilisation (bilateral oophorectomy or hysterectomy)
10. Patients is willing and able to comply with the protocol for the duration of the study including undergoing treatment and scheduled visits and examinations.

Exclusion Criteria:

1. Involvement in the planning and/or conduct of the study (applies to both AstraZeneca staff and/or staff at the study site)
2. Previous enrolment in the present study
3. Participation in another clinical study with an investigational product during the most recent chemotherapy course
4. Any previous treatment with PARP inhibitor, including olaparib
5. Other malignancy within the last 5 years except: adequately treated non-melanoma skin cancer, curatively treated in situ cancer of the cervix, ductal carcinoma in situ (DCIS), Stage 1, grade 1 endometrial carcinoma, or other solid tumours including lymphomas (without bone marrow involvement) curatively treated with no evidence of disease for ≥5 years. Patients with a history of localised triple negative breast cancer may be eligible, provided they completed their adjuvant chemotherapy more than three years prior to registration, and that the patient remains free of recurrent or metastatic disease
6. Resting ECG with QTc > 470 msec on 2 or more time points within a 24 hour period or family history of long QT syndrome
7. Patients receiving any systemic chemotherapy or radiotherapy (except for palliative reasons) within 3 weeks prior to study treatment
8. Concomitant use of known strong CYP3A inhibitors (eg. itraconazole, telithromycin, clarithromycin, protease inhibitors boosted with ritonavir or cobicistat, indinavir, saquinavir, nelfinavir, boceprevir, telaprevir) or moderate CYP3A inhibitors (eg. ciprofloxacin, erythromycin, diltiazem, fluconazole, verapamil). The required washout period prior to starting olaparib is 2 weeks.
9. Concomitant use of known strong (eg. phenobarbital, enzalutamide, phenytoin, rifampicin, rifabutin, rifapentine, carbamazepine, nevirapine and St John's Wort ) or moderate CYP3A inducers (eg. bosentan, efavirenz, modafinil). The required washout period prior to starting olaparib is 5 weeks for enzalutamide or phenobarbital and 3 weeks for other agents.
10. Persistent toxicities (>Common Terminology Criteria for Adverse Event (CTCAE) grade 2) caused by previous cancer therapy, excluding alopecia.
11. Patients with myelodysplastic syndrome/acute myeloid leukaemia or with features suggestive of MDS/AML.
12. Patients with symptomatic uncontrolled brain metastases. A scan to confirm the absence of brain metastases is not required. The patient can receive a stable dose of corticosteroids before and during the study as long as these were started at least 4 weeks prior to treatment. Patients with spinal cord compression unless considered to have received definitive treatment for this and evidence of clinically stable disease for 28 days.
13. Major surgery within 2 weeks of starting study treatment, or patients have not recovered from any effects of any major surgery.
14. Patients considered a poor medical risk due to a serious, uncontrolled medical disorder, non-malignant systemic disease or active, uncontrolled infection. Examples include, but are not limited to, uncontrolled ventricular arrhythmia, recent (within 3 months) myocardial infarction, uncontrolled major seizure disorder, unstable spinal cord compression, superior vena cava syndrome, extensive interstitial bilateral lung disease on High Resolution Computed Tomography (HRCT) scan or any psychiatric disorder that prohibits obtaining informed consent.
15. Patients unable to swallow orally administered medication and patients with gastrointestinal disorders likely to interfere with absorption of the study medication.
16. Breast feeding women.
17. Immunocompromised patients, e.g., patients who are known to be serologically positive for human immunodeficiency virus (HIV).
18. Patients with a known hypersensitivity to olaparib or any of the excipients of the product.
19. Patients with known active hepatitis (i.e. Hepatitis B or C) due to risk of transmitting the infection through blood or other body fluids
20. Previous allogenic bone marrow transplant or double umbilical cord blood transplantation (dUCBT)
21. Whole blood transfusions in the last 120 days prior to entry to the study (packed red blood cells and platelet transfusions are acceptable, for timing refer to inclusion criteria no.6)

Ages: 18 Years to 130 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 229 (Actual)
Dates: Start 2018-05-29 (Actual); Primary Completion 2025-01-27 (Actual); Study Completion 2025-01-27 (Actual)

PRIMARY OUTCOMES:
Time from first dosing date of olaparib to date of disease progression or death from any cause (if this occurs before disease progression) | from first dosing date until objective radiological disease progression by RECIST 1.1, or death from any cause, whichever come first, assessed 45 months.
  Progression free survival (using investigator assessment) according to modified Response Evaluation Criteria In Solid Tumours (RECIST 1.1) of olaparib tablets maintenance monotherapy in platinum sensitive relapsed ovarian cancer patients who are in complete or partial response following platinum based chemotherapy

SECONDARY OUTCOMES:
Time from first dosing date of olaparib to date of disease progression or death from any cause (if this occurs before disease progression) | from first dosing date until objective radiological disease progression by RECIST 1.1, or death from any cause, whichever come first, assessed 45 months.
  Progression free survival (using investigator assessment) according to modified Response Evaluation Criteria In Solid Tumours (RECIST 1.1) of olaparib tablets maintenance monotherapy in BRCA mutated platinum sensitive relapsed ovarian cancer patients who are in complete or partial response following platinum based chemotherapy
Time from first dosing date of olaparib to date of death from any cause | from first dosing date to death, assessed 45 months.
  Assessment of overall survival (OS) of olaparib maintenance monotherapy in platinum sensitive relapsed ovarian cancer patients who are in complete or partial response following platinum based chemotherapy.
Time from first dosing date of olaparib to date of second progression event or death from any cause (if this occurs before second progression event) | from first dosing date to second progression, or death from any cause, whichever come first, assessed 45 months.
  Assessment of time from first dose date to second progression （investigator opinion of progression status）of olaparib maintenance monotherapy in platinum sensitive relapsed ovarian cancer patients who are in complete or partial response following platinum based chemotherapy.
Time from first dosing date of olaparib to date of first subsequent treatment commencement or death from any cause (if this occurs before commencement of first subsequent treatment) | Time from first dosing date of olaparib to date of first subsequent treatment commencement or death from any cause (whichever earlier), assessed 45 months.
  Assessment of time to first subsequent therapy or death (TFST) of olaparib maintenance monotherapy in platinum sensitive relapsed ovarian cancer patients who are in complete or partial response following platinum based chemotherapy.
Time from first dosing date of olaparib to date of second subsequent treatment commencement or death from any cause (if this occurs before commencement of second subsequent treatment) | Time from first dosing date of olaparib to date of second subsequent treatment commencement or death from any cause (whichever earlier), assessed 45 months.
  Assessment of time to second subsequent therapy or death (TSST) of olaparib maintenance monotherapy in platinum sensitive relapsed ovarian cancer patients who are in complete or partial response following platinum based chemotherapy.
Time from first dosing date of olaparib to date of olaparib discontinuation or death from any cause (if this occurs before discontinuation of olaparib maintenance therapy) | Time from first dosing date of olaparib to date of olaparib discontinuation or death from any cause (whichever earlier), assessed 45 months.
  Assessment of time to olaparib discontinuation or death (TDT) of olaparib maintenance monotherapy in platinum sensitive relapsed ovarian cancer patients who are in complete or partial response following platinum based chemotherapy.

OTHER OUTCOMES:
AEs/SAEs | AEs and SAEs collected from informed consent until post treatment 30-day follow-up period, assessed 45 months.
  To assess the safety and tolerability of olaparib maintenance monotherapy in platinum sensitive relapsed ovarian cancer patients
clinical chemistry/haematology parameters. | assessment until post treatment 30-day follow-up period, assessed 45 months.
  To assess the safety and tolerability of olaparib maintenance monotherapy in platinum sensitive relapsed ovarian cancer patients.
Immune-markers PD-L1 expression in tumor tissues | PD-L1 expression in tumor tissues before olaparib treatment.
  To explore biomarkers in tumor tissues predictive of sensitivity/resistance to the treatment of olaparib.
BRCA mutation status in the cell-free DNA from blood samples | at screening (from -28 days to -1 day before baseline)
  To explore biomarkers in blood predictive of sensitivity/resistance to the treatment of olaparib.
other HRR mutation status in the cell-free DNA from blood samples | at screening (from -28 days to -1 day before baseline)
  To explore biomarkers in blood predictive of sensitivity/resistance to the treatment of olaparib.

CONTACTS AND LOCATIONS:
Overall Officials: Ding MA, PhD, Principal Investigator — Tongji Hospital, Tongji Medical College of Huazhong University of Sicence and Technology
Locations (19):
- China (14):
  - Research Site, Beijing
  - Research Site, Changsha
  - Research Site, Chengdu
  - Research Site, Chongqing
  - Research Site, Hangzhou
  - Research Site, Harbin
  - Research Site, Hefei
  - Research Site, Jinan
  - Research Site, Shanghai
  - Research Site, Shenyang
  - Research Site, Tianjin
  - Research Site, Wuhan
  - Research Site, Xi'an
  - Research Site, Zhengzhou
- Malaysia (5):
  - Research Site, Ampang
  - Research Site, Johor Bahru
  - Research Site, Kuala Lumpur
  - Research Site, Kuching
  - Research Site, Putrajaya

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal.
  All request will be evaluated as per the AZ disclosure commitment:
  https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure. Yes, indicates that AZ are accepting requests for IPD, but this does not mean all requests will be shared.
Supporting Information: Study Protocol, SAP
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the deidentified individual patient-level data in an approved sponsored tool . Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home

REFERENCES:
- [Derived] Li H, Peng Z, Zhu J, Zhao W, Huang Y, An R, Zheng H, Qu P, Wang L, Zhou Q, Wang D, Lou G, Wang J, Wang K, Kong B, Xie X, Yin R, Low J, Rozita AM, Sen LC, Meng YC, Kiong KS, Liu J, Liang Z, Lv W, Zhu Y, Hu W, Sun W, Su J, Wang Q, Zang R, Ma D, Gao Q. Exploratory biomarker analysis in the phase III L-MOCA study of olaparib maintenance therapy in patients with platinum-sensitive relapsed ovarian cancer. BMC Med. 2024 May 16;22(1):199. doi: 10.1186/s12916-024-03409-9. PMID 38755585
- [Derived] Gao Q, Zhu J, Zhao W, Huang Y, An R, Zheng H, Qu P, Wang L, Zhou Q, Wang D, Lou G, Wang J, Wang K, Low J, Kong B, Rozita AM, Sen LC, Yin R, Xie X, Liu J, Sun W, Su J, Zhang C, Zang R, Ma D. Olaparib Maintenance Monotherapy in Asian Patients with Platinum-Sensitive Relapsed Ovarian Cancer: Phase III Trial (L-MOCA). Clin Cancer Res. 2022 Jun 1;28(11):2278-2285. doi: 10.1158/1078-0432.CCR-21-3023. PMID 35131903